CLINICAL TRIAL: NCT06940635
Title: Cross-Stroke Therapy Effects With BCI and FES Stimulation: A Pilot Study
Brief Title: Exploratory Study on the Potential Cross-System Effects of BCI-FES Hand Therapy on Dysphagia and Aphasia in Chronic Stroke Patients
Acronym: c-STEPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VASCage GmbH (Other)
Collaborators: g.tec medical engineering GmbH (Industry); Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C_2_BC.4.2_0046_010
Record Dates: First submitted 2025-04-02; First posted 2025-04-23 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Ischaemic Stroke; Hemorrhagic Stroke
Keywords: neurorehabilitation; BCI-FES; chronic stroke; aphasia; dysphagia
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Aphasia; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): 25 BCI-FES therapy sessions over 13 weeks
  Interventions: Device: closed-loop BCI-FES device

INTERVENTIONS:
Device: closed-loop BCI-FES device — Closed-loop neurorehabilitation system that combines EEG-based brain-computer interface technology with functional electrical stimulation (FES) to facilitate neural and motor recovery.

SUMMARY:
The goal of this neurorehabilitation explorative study is to investigate how a closed-loop Brain-Computer Interface Functional Electrical Stimulation (BCI-FES) therapy, used within the intended purpose for hand rehabilitation, may impact swallowing difficulties (dysphagia) and language disorders (aphasia) in post-stroke patients.

DETAILED DESCRIPTION:
Stroke is the leading cause of permanent disability worldwide. Neurorehabilitation (i.e. physical, occupational, and speech/swallowing therapy) is essential for neurological recovery after stroke. According to principles of neuroplasticity and motor learning, key elements are high-intensity training paradigms with task repetition, therapy feedback and cueing modalities. Technical equipment can assist therapists in reaching these aims, for example by facilitating self-training.

One significant technological advancement in this therapeutic field is Brain-Computer Interface (BCI). BCI most commonly uses EEG-signals (i.e. electroencephalography) to capture task related electrical brain activities related to Motor Imagery (MI) translating it for "closed" neurofeedback. Moreover, BCI is frequently coupled with Functional Electrical Stimulation (FES), which stimulates physical movement in the paretic limb while the MI-related tasks are executed. The processed signals are translated into commands to control an external device. The combination of BCI-feedback technology and FES is primarily used to ensure concurrent sensory feedback with motor intention of a goal-based task to restore sensory-motor functions. In the current approach electrical activity related to the MI of upper limb movements is captured and transferred to a corresponding avatar on a computer screen as feedback for the patient.

c-STEPS is designed as a open-label, single-centre, non-controlled, prospective explorative interventional pre-post study. The primary objective of this study is to explore changes in dysphagia or aphasia in stroke patients with arm paresis treated with a closed-loop BCI-FES therapy (used within the intended purpose for hand rehabilitation). Further study objectives are to assess the impact of established treatment protocols on overall independence, disease severity and quality of life related to dysphagia and aphasia, and to investigate simultaneous recovery patterns in hand motor function, dysphagia, and aphasia using a BCI-FES system.

c-STEPS will enroll 10 participants (+2 potential replacements) who are in the chronic post-stroke phase (≥3 months after an ischemic or haemorrhagic stroke). Participants must present with residual arm paresis and either dysphagia (MUCCS-N ≥2) and/or aphasia (AAT ≤3).

Key exclusion criteria include cognitive impairments affecting compliance, brainstem/cerebellar strokes, previous disabling stroke, uncontrolled epilepsy, pacemakers or implanted devices incompatible with FES, severe neglect or anosognosia, and ongoing botulinum toxin treatment. Participants with severe cardiovascular or respiratory conditions (NYHA IV, COPD IV) or other medical risks affecting safety will also be excluded.

The participants will undergo 25 BCI-FES therapy sessions over 13 weeks (twice a week, 45-minute sessions). Throughout the intervention period, interim assessments will be conducted at predefined time points to evaluate treatment progress. A post-treatment assessment will be performed one week after the final therapy session, with additional follow-up assessments at 4 weeks and 26 weeks post-treatment. The overall study duration per participant is 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be aged 18 years or older.
* Post-Stroke Phase: Participants must be within the chronic post-stroke phase (time since ischemic or haemorrhagic stroke greater than 3 months).
* Motor Impairment: Participants must exhibit disabling left or right residual arm paresis ("left/right arm motor drift" part of the NIHSS score ≥1).
* Speech/Swallowing Impairment: Participants must have:

  * Aphasia (AAT-Skala zum Kommunikationsverhalten score ≤3), and/or
  * Dysphagia (MUCCS-N score ≥2).
* Stable Neurological Status: No relevant changes in neurological status in the past 4 weeks (self-reported).
* Motor Function: Participants must be able to raise at least 1 block similar to the ones in Box-and-Block-Test.
* Cognitive Understanding: Participants must be able to understand basic spoken instructions.
* Sitting Tolerance: Participants must be able to maintain a sitting position for at least 60 minutes.
* Willingness to Participate: Participants must be willing to participate in the study and able to understand and sign the informed consent.

Exclusion Criteria:

* Cognitive Impairments: Cognitive impairments that, in the investigator's judgment, could limit understanding of task instructions.
* Stroke Location: Participants with a brainstem and/or cerebellar stroke.
* Previous Stroke: Participants with a previous disabling stroke.
* Hemi-Neglect: Pronounced hemi-neglect at the last documented therapy visit that limits compliance with treatment intervention (investigator's judgment).
* Anosognosia: Pronounced anosognosia at the last documented therapy visit that limits compliance with treatment intervention (investigator's judgment).
* Spasticity: Severe spasticity in the affected limb, resulting in complete rigidity in flexion or extension.
* Seizure Disorders: Participants with uncontrolled epilepsy (investigator's judgement) or epileptic seizure within the last month.
* Intracranial Pressure: Known ongoing elevated intracranial pressure.
* Implanted Medical Devices: Participants with implanted medical devices with contraindication for FES such as pacemakers.
* Metallic Fragments: Participants with implanted metallic fragments in the extremity planned for FES that would limit the use of functional electrical stimulation (FES).
* Unhealed Injuries: Unrecovered fractures or skin/tissue lesions in the FES stimulated extremity.
* Joint Issues: Ossification, contraction, or stiffness of the wrist joint in the FES stimulated extremity that would limit treatment.
* Botulinum Toxin: Participants who received botulinum-toxin treatment within 6 weeks prior to study inclusion and/or for whom botulinum-toxin treatment is planned during the study duration.
* Co-morbidities: The following conditions will exclude participation:

  * Chronic Obstructive Pulmonary Disease (Stage IV).
  * Cardiac insufficiency (NYHA Stage IV).
  * Severe acute infections.
  * Significant circulatory disturbances in the stimulated extremity.
  * Sensory disorders that significantly impair the patient's ability to feel pain or react to unsuitable proprioceptive stimuli.
  * Any other general medical conditions that, in the investigator's judgment, limit the safety or performance of study procedures (investigator's judgement).
* Electrical Stimulation Intolerance: Known inability to tolerate cutaneous electrical stimulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Gugging Swallowing Screen (GUSS) | Baseline, treatment session 16, week 17, week 21 and week 47
  The GUSS is a standardised assessment tool used to evaluate swallowing ability and the risk of aspiration in patients with dysphagia. 4-step clinical assessment; total score ranges from 0 to 20 points. It includes an initial screening followed by assessments of different consistencies of food and drink to determine swallowing safety.
Change in Bielefeld Aphasia Screening Reha (BIAS-R) | Baseline, treatment session 16, week 17, week 21 and week 47
  The BIAS-R is a validated, and standardised assessment tool specifically designed to assess language impairments in aphasic patients in the post-acute stage. It evaluates different aspects of language function such as comprehension, expression, and overall communication ability for different linguistic domains. It is a score-based aphasia screening tool; total score indicates severity of language impairment.

SECONDARY OUTCOMES:
Change in Munich Swallowing Score (MUCCS) | Baseline, week 17, week 21 and week 47
  The MUCCS assesses swallowing function by rating specific criteria related to oral and pharyngeal swallowing phases on two subscales related to saliva swallow (MUCCS-S and oral intake (MUCCS-N). It is a 16-point Likert scale clinical rating.
Change in M.D. Anderson Dysphagia Inventory (M.D.ADI) | Baseline, week 17, week 21 and week 47
  The M.D.ADI evaluates the impact of dysphagia on a patient's quality of life. 20-item, 5-point Likert scale per item. Provides subscale scores (emotional, functional, physical) and a total composite score. Composite Score ranges from 20 (extremely low functioning) to 100 (high functioning).
Change in Communication Outcome after Stroke (COAST) | Baseline, week 17, week 21 and week 47
  The COAST measures the impact of stroke on communication abilities and social participation, focusing on how well individuals are able to interact in everyday situations. The primary caregiver of the study participant will complete this outcome assessment. 2 domains, each item rated on a 5-point Likert scale.
Change in Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | Baseline, week 17, week 21 and week 47
  The FMA-UE is a stroke-specific assessment used to evaluate motor recovery in the upper extremity, focusing on range of motion, coordination, and reflexes. Ordinal 3-point scale per item (0-2); maximum score: 66.
Change in Nine-Hole Peg Test (NHPT) | Baseline, treatment sessions 6, 16 and 21, week 17, week 21 and week 47
  The NHPT measures fine motor skills and dexterity of the upper extremity, particularly focusing on hand function. Performance-based timed test; outcome = time in seconds required to complete the task.
Change in Box-and-Block Test (BBT) | Baseline, week 17, week 21 and week 47
  The BBT is a standardised test used to evaluate gross manual dexterity. It assesses the patient's ability to grasp, lift, and transfer blocks from one side of a box to another. Performance-based test; outcome = number of blocks transferred in 60 seconds.
Change in Scores of Independence for Neurologic and Geriatric Rehabilitation (SINGER) | Baseline, week 17, week 21 and week 47
  The SINGER measures independence in daily activities and is specifically designed for neurological and geriatric rehabilitation settings. Ordinal scale; higher scores reflect greater independence in daily activities during neurorehabilitation.
Change in European Quality of Life 5 Dimensions 3 Level Version (EQ-5D-3L) | Baseline, week 17, week 21 and week 47
  The EQ-5D-3L is a widely used instrument to assess health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 3-level ordinal scale. The EQ-5D-3L also contains a visual analogue scale (VAS) from 0 to 100.
Change in Scale for Measuring Digital Technology Acceptance Adapted for Digital Therapeutic Devices (DTAS-th) | Treatment Sessions 6 and 21, week 17
  The DTAS-th is an adapted instrument originally designed to assess the acceptance of new technologies. The DTAS-th emphasizes two key dimensions: perceived usefulness, which refers to the therapists' view of how effective the treatment method is in improving patient outcomes, and perceived ease of use, which captures how user-friendly and practical the method is from the therapists' perspective. 13-item questionnaire based on the Technology Acceptance Model (TAM). Each item is rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knoflach, Assoc.-Prof., Principal Investigator — Medical University of Innsbruck
Locations (1):
- Department for Neurology, Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No